CLINICAL TRIAL: NCT03073382
Title: Risk Factors Associated With Spontaneous Preterm Delivery Status Post Open Fetal Myelomeningocele Repair
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: St. Louis University (Other)
Responsible Party: Sponsor
Other Study IDs: 26891
Record Dates: First submitted 2017-02-01; First posted 2017-03-08 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Myelomeningocele
MeSH Terms: conditions — Meningomyelocele

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Chart review — This is a chart review of all patients who have underwent open prenatal repair of fetal myelomeningocele. Although prenatal repair is associated with improved neurologic outcomes and a decreased need for cerebrospinal fluid shunting after birth, one of the major risks is preterm delivery. This study is intended to identify maternal, fetal or intraoperative risk factors associated with preterm delivery.

SUMMARY:
This is a chart review of all patients who have underwent open prenatal repair of fetal myelomeningocele. Although prenatal repair is associated with improved neurologic outcomes and a decreased need for cerebrospinal fluid shunting after birth, one of the major risks is preterm delivery. This study is intended to identify maternal, fetal or intraoperative risk factors associated with preterm delivery.

DETAILED DESCRIPTION:
Myelomeningocele encompasses the most common form of spina bifida. The incidence ranges from 2.73-3.80 per 10,000 births in the United States. The extent of neurologic sequela is correlated with the level of the lesion but frequently involves a spectrum of motor dysfunction including paralysis of the lower extremities, contractures in addition to lack of bladder and bowel control. These result in significant lifestyle limitations for survivors. Additionally, hydrocephalus, brainstem herniation and Chiari II malformations are commonly noted. Ventriculoperitoneal shunts are commonly placed in childhood to redirect cerebrospinal fluid and can require revisions later in life.

The Management of Myelomeningocele Study (MOMS) trial revolutionized management of fetuses with myelomeningoceles by demonstrating that prenatal compared to standard postnatal repair resulted in decreased need for cerebrospinal fluid shunts and improved motor function at thirty months. As a result, various centers around the United States began offering prenatal repair to patients less than twenty-six weeks gestation with prespecified maternal and fetal characteristics.

Prenatal repair is not without risk to both the mother and the fetus. The mother must undergo a laparotomy and accept the risks involved with any intraabdominal surgery including bleeding, infection, adhesion formation and damage to nearby organs. Unique to this procedure, a hysterotomy is typically created in the active segment of the uterus to allow for sufficient exposure of the fetal lesion. Like those women who undergo classical Cesarean sections, these patients must undergo Cesarean sections around 37 weeks gestation for all future pregnancies secondary to concern of uterine dehiscence in the setting of labor. This has major implications for the mother's future childbearing potential, as the number of previous Cesarean sections increases the risk of intraoperative complications and invasive placentation in subsequent pregnancies. A fetoscopic approach has reemerged in the United States as an alternative to the aforementioned open approach and is currently under further investigation.

Intraoperative fetal distress has been reported and can lead to loss of the pregnancy. Additionally, fetal surgery carries the risks of spontaneous preterm birth and preterm premature rupture of membranes, which subject the fetus to the morbidity of prematurity. This risk of spontaneous preterm delivery is one of the more common and significant drawbacks to the procedure and represents a major hurdle to overcome. In the MOMS trial, 46% of those in the study group compared to 8% in the postnatal repair group experienced spontaneous rupture of membranes. Thirty-eight percent of prenatal repair versus 14% of postnatal repair patients went into spontaneous labor prior to scheduled delivery. The average gestational age at birth was 34 weeks for the prenatal surgery group and 37 weeks for the postnatal surgery group. In another study following the MOMS trial, 100 patient underwent prenatal repair with a reported 32.3% rate of preterm premature rupture of membranes(PPROM) and 37.5% rate of preterm labor. Also reported a modified surgical approach to the hysterotomy and closure among 43 patients and found a 22% rate of PPROM. Thirty-nine percent delivered at 37 weeks or later compared with 21% of the MOMS cohort.

Although the increased risk of preterm delivery is reported, little is known regarding risk factors associated with preterm delivery following this procedure. Soni et al. found that chorioamniotic membrane separation was a risk factor for subsequent PPROM. No studies have been published that assess risk factors for all spontaneous preterm deliveries including both preterm labor and PPROM. The objective of this study is to determine if any maternal, fetal or intraoperative factors can be identified that increase the risk of spontaneous preterm delivery in patients who undergo prenatal open myelomeningocele repair. With the identification of such factors, counseling of the patient and potentially patient selection could be refined in the future.

ELIGIBILITY:
Inclusion Criteria:

* chart review of all patients who have underwent open prenatal repair of fetal myelomeningocele.

Exclusion Criteria:

* excluded if delivery information is unavailable.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients who underwent open fetal myelomeningocele repair Ethnicity: Any
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2017-05-26 (Actual)

PRIMARY OUTCOMES:
The number of spontaneous preterm delivery | 1 year
  Although prenatal repair is associated with improved neurologic outcomes and a decreased need for cerebrospinal fluid shunting after birth, one of the major risks is preterm delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Heather H Said, MD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No